CLINICAL TRIAL: NCT03024294
Title: Care Pathway for Patients Undergoing VATS Lobectomy or Segmentectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Scott J Swanson, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016P002308
Record Dates: First submitted 2017-01-06; First posted 2017-01-18 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: VATS Lobectomy; VATS Segmentectomy; Care Pathway; Lung Nodule
MeSH Terms: interventions — Mastectomy, Segmental

ARMS (1):
- Patients undergoing VATS lobectomy or segmentectomy (Other): Patients undergoing VATS lobectomy or segmentectomy performed by one of the surgeons in the Division of Thoracic Surgery who are then placed on this specific post-operative care pathway to determine the rate of discharge of these patients by post-operative day (POD) three.
  Interventions: Other: Post-operative care pathway for patients undergoing VATS lobectomy or segmentectomy

INTERVENTIONS:
Other: Post-operative care pathway for patients undergoing VATS lobectomy or segmentectomy — To place participants on this specific post-operative care pathway upon the completion of their VATS surgery to determine the discharge rate by midnight on post-operative day (POD) three.

SUMMARY:
The goal of this study is to create a unified SOP for care of subjects undergoing VATS lobectomy and segmentectomy by members of the Division of Thoracic Surgery. Other academic centers have created standardized algorithms for the care of their subjects and this enables the centers to determine which subjects can be placed on an accelerated pathway to discharge and which cannot. Some of these SOPS dictate uniform treatment algorithms with reduction in what may be unnecessary tests to simplify patient care and likely accelerate them towards safe and more timely discharge from the hospital.

DETAILED DESCRIPTION:
This is a prospective, study to develop, test, fine-tune and refine an SOP for the post-operative care for patients who undergo a VATS lobectomy or segmentectomy performed by one of the surgeons in The Division of Thoracic Surgery. This study will be conducted in two phases. Phase 1 will be focused on early feasibility of the SOP and this will be done by enrolling 50 participants among the subgroup of Thoracic VATS Surgeons who participate. An analysis will take place upon the completion of the phase 1 to look at the percentage of participants who were able to be discharged on or prior to POD 3. Upon this analysis, modifications across all areas of the care pathway will be evaluated and altered if deemed necessary by the PI and other members of the study team. This analysis will drive any modifications needed that will be incorporated into the phase II design prior to its implementation. The treating Thoracic Surgeon for each patient will follow the SOP as it is outlined and the steps the post-operative team will follow will be dependent on which phase the participant is enrolled too. Data will be collected for each participant starting just prior to the VATS operation and continue through the discharge and conclude once the participants have reached their 90-day post-discharge date. Upon discharge from the hospital the participant will enter the follow-up period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age ≥ 18 years
* Subjects planned to undergo a VATS lobectomy or segmentectomy procedure for lung nodules

Exclusion Criteria:

* Subjects who cannot undergo VATS surgery
* Subjects undergoing any kind of resection in addition to VATS Lobectomy or Segmentectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate feasibility of this SOP in two phases. The primary objective of phase 1 is to determine the POD 3 rate, defined as proportion of patients who are discharged by midnight on POD 3. | From date of consent until midnight of post op day 3
The primary objective of phase II is to further evaluate this SOP. The study team will also have the opportunity to refine and fine tune this SOP between phase I and phase II. | From date of consent until midnight of post op day 3

CONTACTS AND LOCATIONS:
Overall Officials: Scott Swanson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States